CLINICAL TRIAL: NCT06742229
Title: Prospective Clinical Data Collection for Developing Machine Learning-assisted Obstetric Ultrasound (MOBUS) Screening Algorithms
Brief Title: Clinical Data Collection for Obstetric Ultrasound Algorithms
Acronym: MOBUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caption Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAP-MOBUS-24-02
Record Dates: First submitted 2024-12-10; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy
Keywords: Obstetrics; Gynecology; Artificial Intelligence; Machine Learning

STUDY DESIGN:
Intervention Model Description: Two groups- Group 1 Pregnant and Group 2 Non Pregnant. From Group 1-Pregnant group we will obtain their standard of care scans along with the research scan whereas Non pregnant group will have only research scans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1: Pregnant Subjects (Other): This group is for pregnant subjects. They will have two ultrasound scans performed- One will be the standard of care ultrasound scan and the other will be research scan
  Interventions: Device: Research Ultrasound scan
- Group 2- Non pregnant Subjects (Other): This group is for non-pregnant subjects. They will have one ultrasound scan performed- it will be the research scan
  Interventions: Device: Research Ultrasound scan

INTERVENTIONS:
Device: Research Ultrasound scan — Both the study groups will be asked to undergo a research scan performed by an FDA approved ultrasound device

SUMMARY:
The goal of this clinical trial is to

* Collect ultrasound data from pregnant and non-pregnant individuals presenting to multiple study sites.
* Use the collected data and ultrasound images to train and validate Artificial intelligence algorithms developed by the Sponsor

Consented participants will be asked to take part in a research ultrasound scan

DETAILED DESCRIPTION:
In this study pregnant and no pregnant subjects will be recruited from Obstetrics and Gynecology clinics/hospitals or from Maternal and Fetal Medicine centers. The pregnant subjects will be in Group 1 and non pregnant subjects will be in Group 2. Pregnant subjects are only recruited if they are scheduled for an obstetric standard of care scan . Both the group will undergo research scan, which is a sweep protocol using handheld FDA approved ultrasound device like Vscan. Patient chart history (no PHI), standard of care scan ultrasound images (no PHI), and research scan ultrasound images (no PHI) would be obtained from Group 1 subjects. Patient history (no PHI), research ultrasound images (no PHI) would be obtained from Group 2 subjects The data collected from this study will be used by the sponsor to develop algorithms for screening various fetal health parameters such as gestational age, placenta location, fetal heart rate, number of fetuses, fetal positions etc

Th

ELIGIBILITY:
Inclusion Criteria:

Pregnant group (Group 1)

1. Participants aged 18 years or older at time of consent.
2. Participants with confirmed pregnancy (positive HCG urine test strip and/or a documented obstetric ultrasound scan.
3. Participants who are scheduled for or referred for a standard-of-care clinical obstetric ultrasound examination.
4. Participants who provide written consent.

Non-pregnant group (Group 2)

1. Participants aged 18 years or older at time of consent.
2. Participants who are not actively pregnant (confirmed using an HCG urine test strip).
3. Participants who provide written informed consent.

Exclusion Criteria:

- 1. Participants for whom participating in this study would delay or compromise care in any way.

2. Participants who are not able to understand or provide written consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Research sweep Ultrasound Images (Vscan ) from the participants will be assessed for quality of images and comparing with patient chart history | 9 months
  All the participant's research ultrasound image will be obtained. This image will be checked for image quality on various stages of pregnancy as well as for non pregnant subjects. These images will be used to develop algorithms for measuring gestational age, placenta location etc.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No